CLINICAL TRIAL: NCT00442689
Title: Metabolic Syndrome in PCOS: Precursors and Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andrea Dunaif, Charles F Kettering Professor of Endocrinology & Metabolism Vice Chair for Research, Department of Medicine Northwestern University, Feinberg School of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: DK73411; R01DK073411 (NIH)
Record Dates: First submitted 2007-02-05; First posted 2007-03-02 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Polycystic Ovary Syndrome; Metabolic Syndrome
Keywords: Polycystic Ovary Syndrome; Metabolic Syndrome; PCOS; overweight; infertility; Insulin Resistance; menstrual cycle
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Syndrome; Overweight; Infertility; Insulin Resistance | interventions — Flutamide; Ethinyl Estradiol; drospirenone; drospirenone and ethinyl estradiol combination; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): oral contraceptive (35 mg ethinyl estradiol)
  Interventions: Drug: ethinyl estradiol 35 mcg and drospirenone 3 mg
- 2 (Experimental): Flutamide 250 mg twice daily
  Interventions: Drug: flutamide
- 3 (Placebo Comparator): Placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: flutamide — 250 mg twice daily
  Other Names: Eulexin
  Arms: 2
Drug: ethinyl estradiol 35 mcg and drospirenone 3 mg — one active pill per day for three weeks and then 1 sugar pill per day for one week
  Other Names: Yasmin
  Arms: 1
Other: placebo
  Other Names: sugar pill
  Arms: 3

SUMMARY:
The purpose of this study is to investigate the metabolic effects of anti-androgens and oral contraceptive pills (OCPs), compared with placebo, in the treatment of women with PCOS. We hypothesized that controlling elevated androgen levels with either anti-androgens or OCPs would produce improvement in metabolic markers in PCOS women and would reduce their long term metabolic risk.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is one of the most common conditions of young women, and it is frequently associated with insulin resistance or metabolic syndrome (MBS). In addition, affected women have significantly elevated mean low-density lipoprotein (LDL) levels and an increased prevalence of at risk LDL levels, independent of obesity. We are directly testing the role of androgens in the metabolic abnormalities in PCOS by examining the impact of direct androgen receptor blockade by anti-androgen medications and indirect suppression of androgen production through suppression of leutinizing hormone (LH) with oral contraceptive pills (OCPs), compared with placebo, on visceral adiposity, circulating LDL levels, insulin secretion and sensitivity as measured by frequently-sampled IV glucose tolerance tests (FSIGT) and oral glucose tolerance tests (OGTT), resting energy expenditure, and maximal aerobic capacity measurement.

Note: Originally there were 2 additional study arm, Metformin only and Metformin + Flutamide. These study arms were ultimately eliminated and were not included in analysis of baseline characteristics or endpoints.

ELIGIBILITY:
Inclusion Criteria:

* 6 periods or fewer per year
* Overweight
* All ethnicities

Exclusion Criteria:

* Diabetes
* Heart Disease
* Chronic illness
* Regular Smokers
* Current use of Birth Control Pills, Patch, Ring, Depo

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2006-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Dunaif, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Diamanti-Kandarakis E, Mitrakou A, Raptis S, Tolis G, Duleba AJ. The effect of a pure antiandrogen receptor blocker, flutamide, on the lipid profile in the polycystic ovary syndrome. J Clin Endocrinol Metab. 1998 Aug;83(8):2699-705. doi: 10.1210/jcem.83.8.5041. PMID 9709934
- [Background] Gambineri A, Patton L, Vaccina A, Cacciari M, Morselli-Labate AM, Cavazza C, Pagotto U, Pasquali R. Treatment with flutamide, metformin, and their combination added to a hypocaloric diet in overweight-obese women with polycystic ovary syndrome: a randomized, 12-month, placebo-controlled study. J Clin Endocrinol Metab. 2006 Oct;91(10):3970-80. doi: 10.1210/jc.2005-2250. Epub 2006 Jul 25. PMID 16868063
- [Background] Gambineri A, Pelusi C, Genghini S, Morselli-Labate AM, Cacciari M, Pagotto U, Pasquali R. Effect of flutamide and metformin administered alone or in combination in dieting obese women with polycystic ovary syndrome. Clin Endocrinol (Oxf). 2004 Feb;60(2):241-9. doi: 10.1111/j.1365-2265.2004.01973.x. PMID 14725687
- [Background] Urbanek M, Sam S, Legro RS, Dunaif A. Identification of a polycystic ovary syndrome susceptibility variant in fibrillin-3 and association with a metabolic phenotype. J Clin Endocrinol Metab. 2007 Nov;92(11):4191-8. doi: 10.1210/jc.2007-0761. Epub 2007 Sep 4. PMID 17785364

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 97 total subjects enrolled. Prior to randomization, 16 subjects were excluded or dropped out, leaving 81 active subjects. Early in the study, 2 of the 5 study arms were discontinued: participants receiving Metformin only (8 subjects) and those receiving Metformin + Flutamide (6 subjects) - leaving 67 subjects whose data were analyzed
Groups:
- Oral Contraceptive - 1: Oral contraceptive (containing 35mcg of ethinyl estradiol and 3mg of drospirenone)
  Oral contraceptive: one active pill per day for three weeks and then 1 sugar pill per day for one week
- Flutamide - 2: Flutamide
  Flutamide: 250 mg twice daily
- Placebo - 3: Placebo only
Period: Overall Study
Arm/Group | Oral Contraceptive - 1 | Flutamide - 2 | Placebo - 3
Started | 21 | 24 | 22
Completed | 11 | 13 | 13
Not Completed | 10 | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Oral Contraceptive - 1: Oral contraceptive (containing 35mcg of ethinyl estradiol and 3mg of drospirenone)
- Placebo - 3: Placebo
- Total: Total of all reporting groups
Arm/Group | Oral Contraceptive - 1 | Flutamide - 2 | Placebo - 3 | Total
Number analyzed (Participants) | 21 | 24 | 22 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (4) | 28 (4) | 28 (5) | 28 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 22 | 67
  Male | 0 | 0 | 0 | 0
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 37.1 (5.5) | 40.1 (5.6) | 40.0 (6.7) | 39.3 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Low-density Lipoprotein (LDL) Levels Over the Study Period
Description: Change in low-density lipoprotein (LDL) levels over the study period (LDL level at study endpoint - baseline LDL level)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Contraceptive - 1 | Flutamide - 2 | Placebo - 3
Number analyzed (Participants) | 11 | 13 | 13
mg/dL | -6 (17) | -9 (14) | -7 (17)

2. Primary Outcome: Change in High-density Lipoprotein (HDL) Levels During Study Period
Description: Change in high-density lipoprotein (HDL) levels during study period (HDL level at study endpoint - baseline HDL)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Oral Contraceptive - 1 | Flutamide - 2 | Placebo - 3
Number analyzed (Participants) | 11 | 13 | 13
mg/dL | 6 (4) | -5 (7) | -2 (5)

3. Primary Outcome: Change in Visceral Adipose Tissue (VAT) Volume as Measured by MRI
Description: Change in visceral adipose tissue (VAT) volume as measured by MRI (VAT at study endpoint - baseline VAT)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Oral Contraceptive - 1 | Flutamide - 2 | Placebo - 3
Number analyzed (Participants) | 11 | 13 | 13
L | -0.1 (0.3) | -0.1 (0.6) | 0.1 (0.6)

4. Primary Outcome: Change in Fat Percentage as Measured by Dual-energy X-ray Absorptiometry (DEXA) Scan Over the Study Period
Description: Change in fat percentage as measured by DEXA scan over the study period (Fat percentage at study endpoint - baseline fat percentage)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of body mass
Arm/Group | Oral Contraceptive - 1 | Flutamide - 2 | Placebo - 3
Number analyzed (Participants) | 11 | 13 | 13
percentage of body mass | 0.4 (1.5) | -1.9 (3.9) | -1.9 (2.3)

5. Primary Outcome: Change in Disposition Index
Description: Change in disposition index (DI, insulin secretion corrected for insulin secretion) as measured by frequently-sampled IV glucose tolerance test (DI at study endpoint - baseline DI)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: min^-1
Arm/Group | Oral Contraceptive - 1 | Flutamide - 2 | Placebo - 3
Number analyzed (Participants) | 11 | 13 | 13
min^-1 | 1653 (6008) | 194 (1424) | -184 (825)

6. Primary Outcome: Change in Resting Energy Expenditure (REE) Over the Study Period
Description: Change in resting energy expenditure (REE) over the study period (REE at study endpoint - baseline REE)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Kcal/day
Arm/Group | Oral Contraceptive - 1 | Flutamide - 2 | Placebo - 3
Number analyzed (Participants) | 11 | 13 | 13
Kcal/day | 7 (209) | -79 (239) | -88 (203)

7. Primary Outcome: Change in Maximal Aerobic Exercise Capacity (VO2 Max) Over the Study Period
Description: Change in maximal aerobic exercise capacity (VO2 max) over the study period (VO2 max at study endpoint - baseline VO2 max)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Oral Contraceptive - 1 | Flutamide - 2 | Placebo - 3
Number analyzed (Participants) | 11 | 13 | 13
L/min | -0.5 (6.5) | -1.6 (4.4) | 1.1 (4.9)

ADVERSE EVENTS:
Time Frame: 6 months - adverse event data collected over the study period.
Arm/Group | Oral Contraceptive - 1 | Flutamide - 2 | Placebo - 3
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 1/21 | 4/24 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Contraceptive - 1 (N=21) | Flutamide - 2 (N=24) | Placebo - 3 (N=22)
Abnormal LFTs (Hepatobiliary disorders) | 1 (1) | 4 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
Please note there were 2 additional arms at the start of the study: Metformin alone (n=8) and Metformin+Flutamide (n=6), which were discontinued. These arms are therefore not included in these results data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No